CLINICAL TRIAL: NCT06881394
Title: A Pilot, Open-Label, Single Site Study Evaluating the Safety and Efficacy of Topical Cyanoacrylate Antiperspirant in Adults With Palmar Hyperhidrosis
Brief Title: A Polymer Film Device to Treat Excessive Palmar Sweating
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miller Biosciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCAAP-PH
Record Dates: First submitted 2025-02-26; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Palmar Hyperhidrosis
Keywords: palmar hyperhidrosis; polymer film; gravimetric sweat assessment; grip function; hyperhidrosis disease severity scale; topical

STUDY DESIGN:
Intervention Model Description: The study is a single group interventional study model where all participants receive the same in the study arm, and no control group is used. Participants are not randomly assigned to the treatment group but selected based on symptom severity (i.e., their hyperhidrosis disease severity score assess by a clinician). Data on the participants' outcomes will be collected before and after using the device to assess its efficacy and safety. This study model is sufficient to demonstrate device feasibility and assess the safety and usability of a new device in a small study group. The primary and secondary endpoints to be measured are quantitative and will directly assess the device ability to reduce participant including sweat levels and grip function. Robust data collection methods will be implemented to minimize bias and ensure the data is reproducible and informative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Topical TCA treatment once or twice daily (Experimental): Participants with HDSS of 3-4 receiving topical polymer treatment once or twice daily for one week
  Interventions: Device: Polymer Skin Barrier

INTERVENTIONS:
Device: Polymer Skin Barrier — A cyanoacrylate polymer will be applied topically once or twice a day to the palmar surface of hands to prevent perspiration

SUMMARY:
Perspiration or sweating is a normal physiological response to increased body temperature, environmental heat and humidity, emotions, nervousness, or physical exertion. Perspiration occurs when sweat is secreted from sweat glands, travels through sweat ducts and exits sweat pores to coat the skin's surface. The evaporation of sweat from the skin dissipates heat and is the primary thermoregulatory mechanism used by humans and primates. Excessive sweating beyond what is required for maintaining body temperature homeostasis is termed hyperhidrosis. Primary hyperhidrosis is idiopathic affecting the palmar, plantar, axillary, or craniofacial regions bilaterally, while secondary hyperhidrosis is less common and is often a side effect of medication or an underlying pathology. Primary hyperhidrosis may affect up to 4.8% of the US population, yet it is widely underreported and undertreated. Hyperhidrosis can negatively impact daily activities, cause significant stress, limit social interactions, and reduce the quality of life for patients. In particular, excessive palmar sweating interferes with professional activities (e.g., shaking hands, working with tools, or wearing exam gloves) and degrades sports performance.

Hyperhidrosis (HH) is especially difficult to treat on the hands and feet, with clinical care beginning with prescription strength topical aluminum chloride hexahydrate antiperspirants such as DrySol or Secret Clinical, and OTC products (e.g., Carpe). However, prescription strength aluminum chloride antiperspirants are often ineffective, can be irritating and leave a residue that degrades skin texture and grip. Currently, iontophoresis is the only medical device approved for treating palmar and plantar HH, but these devices are expensive (~$1,500), uncomfortable to use and are time consuming (30 minutes sessions, 3-4 times a week for several months). Oral anticholinergic medicines such as oxybutynin are often prescribed but they have unwanted side effects including blurred vision, dry mouth, and headache. Topical anticholinergic wipes have shown promise, but they are expensive, take weeks to relieve symptoms and have unpleasant side effects in >18% of patients. Finally, invasive procedures such as Botox™ injections and endoscopic thoracic sympathectomy are used to treat the most severe palmar/plantar HH cases but these treatments are expensive, invasive, painful and can have significant adverse effects including persistent muscle weakness and compensatory sweating. Thus, a high unmet need exists for topical treatments that are fast-acting, safe, and effective.

Cyanoacrylate (CA) tissue adhesives have been used for decades to close wounds, stop bleeding, and prevent infection. CA tissue adhesives bond to the skin through Michael's addition reactions to tissue amines, forming durable but flexible films. Despite CA being used for various medical applications, no CA-based antiperspirants are currently clinically approved or commercially available.

Topical cyanoacrylate (TCA) is based on medical grade cyanoacrylate adhesives with decades of demonstrated safety clinical applications. TCA is cheap to produce which will improve affordability and treatment adoption. In addition, prototypical TCA formulations eliminate surface moisture within seconds and occlude eccrine sweat pores, anticipating a strong antiperspirant effect compared to current treatments which typically reduce sweating with variable efficacy.

TCA is innovative because it is fast acting (acts within seconds) and does not degrade the surface of the skin or grip function. Current hyperhidrosis treatments typically require days to weeks to achieve clinical results, have a variety of undesirable side effects, and can negatively affect the surface feel of the skin. Aside from topical antiperspirants, Botox injections and anticholinergic agents are the only drugs approved by the FDA for treating hyperhidrosis. Due to their rapid polymerization and strong adhesion and low toxicity, n-Butyl and 2-Octly cyanoacrylate are widely used in thoracic, gastrointestinal, neurologic, cardiovascular, ophthalmologic, and vascular surgery. Although n-Butyl and 2-Octyl cyanoacrylate are considered safe, allergic contact dermatitis can occur after surgical wounds closure at an incident rate of 2.7% for 2-Octyl cyanoacrylate and 2.2% for n-Butyl cyanoacrylate, but risks are presumably lower for topical application on intact glabrous skin. Thus, a significant unmet need exists for fast-acting, cheap, effective, and safe treatments that leave the skin with a desirable surface feel and improve grip security.

In this pilot study described in this proposal, investigators will evaluate the safety and efficacy of a topical application of generic cyanoacrylate (TCA, equivalent to FDA cleared GluStich® medical adhesive or Marathon No Sting Liquid Skin Protectant) to inhibit palmar perspiration.

DETAILED DESCRIPTION:
Protocol TCAAP-PH will investigate TCA use in participants with palmar hyperhidrosis. This is a pilot, open-label, single site study designed to evaluate the safety and efficacy of TCA in participants 18 years of age and older. The study will have a maximum study duration of 4 weeks. This includes screening/baseline, a 1-week treatment period, and a 4 week follow up phone call and exit survey. A total of approximately 30 participants will be enrolled in this study. At the inception of the trial, the age of participants will be 18 years of age or older.

Screening/Baseline will occur the same day to confirm the selection criteria for the study are met. Qualified participants in TCAAP-PH will be selected to receive TCA at this visit. Participants will administer TCA to the affected areas of the palms/fingers daily throughout the treatment period.

This study is being conducted to evaluate the short-term safety and efficacy of TCA dosed up to 1 week of treatment duration. In addition to safety, another objective of this study is to evaluate short-term efficacy in this population. To evaluate the efficacy, response will be assessed based on the hyperhidrosis disease severity scale (HDSS), an instrument that is widely used to assess the severity of palmar hyperhidrosis by the subject that best reflects his or her experience with sweating of the specified body area. Participants are asked "How would you rate the severity of your hyperhidrosis?" (1) My sweating is never noticeable and never interferes with my daily activities (2) My sweating is tolerable but sometimes interferes with my daily activities (3) My sweating is barely tolerable and frequently interferes with my daily activities (4) My sweating is intolerable and always interferes with my daily activities. A score of 3 or 4 indicates severe hyperhidrosis. A score of 1 or 2 indicates mild or moderate hyperhidrosis. A 1-point improvement in HDSS score has been associated with a 50% reduction in sweat production and a 2-point improvement with an 80% reduction. This tool has been well accepted and used in multiple palmar hyperhidrosis clinical trials as a reliable and reproducible measure of palmar hyperhidrosis severity. In addition, gravimetric sweat production and grip strength measurements will be used to assess the short-term efficacy in this population. The total sample size for the study is estimated to be approximately 30 participants.

The TCAAP-PH treatment protocol that is being administered to the study intervention group has been used for other indications (e.g. extraoral wound closures and skin protectants) with minimal risk to patients. Due to the low risk profile of cyanoacrylate, the use of this agent for palmar hyperhidrosis will be evaluated with no significant concern regarding the dosage that will be applied to the affected areas. Dosage is 100 µL once per day, which is sufficient to cover the palmar and phalangeal surface of both hands when properly applied. The solution will be applied in the morning after subjects complete their morning meal and washing routine.

The end of the study is defined as the date of the last visit of the last participant in the study. The date of the last visit will be considered the Week 4 phone call.

ELIGIBILITY:
Inclusion Criteria: Participants must meet all of the following criteria to be eligible for study participation:

1. Signed informed consent.
2. Age ≥ 18 years.
3. Willing to comply with the protocol.
4. Male or non-pregnant (negative urine pregnancy test in female subjects of child-bearing potential), non-lactating females.
5. Primary palmar hyperhidrosis for at least 6 months duration.
6. Average sweat severity score of ≥ 3 at Baseline. Subjects must complete at least 4 days of the sweat severity NRS within 7 days of the Baseline visit.
7. HDSS of 3 or 4 at Baseline.
8. If female and of childbearing potential, subject must be willing to use an accepted method of birth control during study participation and for 30 days after the last study drug application. Females are considered to be of childbearing potential unless surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation), have been diagnosed as infertile, have same gender sex partner, are pre-menarche or are post-menopausal for at least 1 year. Hormonal contraception exclusively for study participation may be prohibited for minor female subjects according to local law and medical practice. Acceptable methods of birth control include: abstinence, oral contraceptives, contraceptive patches/implants; injectable contraceptives, double barrier methods (e.g., condom and spermicide) or an intra-uterine device (IUD). Birth control methods must have been stable/unchanged for 12 weeks prior to baseline and must remain unchanged during study participation.
9. If male, is vasectomized or agrees to use an accepted method of birth control with a female partner during study participation and for 7 days after the last study drug application.

   -

Exclusion Criteria: Participants meeting any of the following criteria are not eligible for study participation:

1. Subjects who have taken or are currently taking Qbrexza (glycopyrronium) 2.4% within 4 weeks of baseline
2. Prior surgical procedure for hyperhidrosis.
3. Iontophoresis for the palms within 4 weeks of Baseline.
4. Treatment with botulinum toxin (e.g., Botox) for palmar hyperhidrosis within 6 months of Baseline.
5. Subjects who are actively participating in an experimental therapy study or who received experimental therapy within 30 days or 5 half-lives (whichever is longer) of the Baseline Visit.
6. Subjects who have had a change in a regimen of psychotherapeutic medication (change in drug, dose, frequency) or who have started a psychoactive medication within two months of Baseline visit.
7. Treatment with medications having systemic anticholinergic activity, centrally acting alpha-2 adrenergic agonists (e.g., clonidine, guanabenz, methyl dopa), or beta-blockers within 4 weeks of the Baseline visit unless dosing has been stable for at least 4 months prior to Baseline and is not expected to change over the course of the study (inhaled anti-cholinergic drugs or beta agonists are allowed).
8. Intravenous (IV), oral, or topical glycopyrrolate treatment or any systemic treatment with an anticholinergic medication such as atropine, belladonna, scopolamine, clindinium or hyoscyamine within 4 weeks prior to Baseline.
9. Current pregnancy or lactation.
10. Open wounds or inflammatory lesions on the hands or, any condition that may alter the barrier function of the skin on the hands.
11. Secondary palmar hyperhidrosis or presence of a condition that may cause secondary hyperhidrosis (e.g., lymphoma, malaria, severe anxiety not controlled by medication, carcinoid syndrome, substance abuse, hyperthyroidism).
12. Screening clinical chemistry or hematology laboratory (if medically necessary) value that is considered clinically significant, in the opinion of the Investigator.
13. Known history of Sjogren's syndrome or Sicca syndrome.
14. History of glaucoma, inflammatory bowel disease, toxic megacolon, active febrile illness, paralytic ileus, unstable cardiovascular status in acute hemorrhage, severe ulcerative colitis, toxic megacolon complicating ulcerative colitis or myasthenia gravis.
15. History or presence of ventricular arrhythmias, atrial fibrillation, atrial flutter. History of other supraventricular tachycardia with a ventricular rate greater than 100 (other than sinus tachycardia).
16. Subjects who are a poor medical risk because of other systemic diseases or active uncontrolled infections, or any other condition which, in the judgment of the Investigator, would put the subject at unacceptable risk for participation in the study.
17. Subjects that have a known or suspected allergy to cyanoacrylates.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Hand sweating severity score | 7 days
  Participants will be assessed for a mean change in hand sweating severity score from Baseline to Day 1 and Day 7 post-treatment. Participants are asked "How would you rate the severity of your hyperhidrosis?" (1) My sweating is never noticeable and never interferes with my daily activities (2) My sweating is tolerable but sometimes interferes with my daily activities (3) My sweating is barely tolerable and frequently interferes with my daily activities (4) My sweating is intolerable and always interferes with my daily activities. A score of 3 or 4 indicates severe hyperhidrosis. A score of 1 or 2 indicates mild or moderate hyperhidrosis. A 1-point improvement in HDSS score has been associated with a 50% reduction in sweat production and a 2-point improvement with an 80% reduction. This tool has been well accepted and used in multiple palmar hyperhidrosis clinical trials as a reliable and reproducible measure of palmar hyperhidrosis severity.
Gravimetric assessment of sweat production | 7 days
  Palmar sweat production in participants will be assessed gravimetrically to measure the mean absolute change in sweat production from baseline to Day 1 and Day 7 post-treatment
Grip function assessment | 7 days
  Participant grip security (force before slippage) will be measured using a hand held dynamometer at baseline and at Day 1 and Day 7 post-treatment

SECONDARY OUTCOMES:
Proportion of subjects with improvement in hand sweating severity score | 7 days
  Proportion of participants who at 1 week have a ≥3-point improvement in mean hand sweating severity score or a ≥2-grade improvement in HDSS from baseline.

OTHER OUTCOMES:
Quality of Life Improvement | 4 weeks
  Participant self-evaluation survey to assess treatment impact on quality of life:
  Q1: Have you experienced itching, pain, redness, swelling or other signs of irritation at the TCA product application site on the hands? If yes, please explain.
  Q2: How effective was the product treatment at reducing perspiration on your hands during the trial?
  1-Not at all, 2-Somewhat, 3-Moderately, 4-Very, 5-Extremely effective Q3: Did TCA have a positive impact on your social, recreational, or professional activities? If so, which activities and how? Q4: How easy was it to apply the product to your hands during the trial?
  1-Not at all, 2-Somewhat, 3-Moderately, 4-Very, 5-Extremely easy Q5: If you tried other palmar hyperhidrosis treatments, how did the TCA product compare?
  1-Worse, 2-Slightly worse, 3-The same, 4-Better, 5-Much better Q6: Do you have any suggestions or feedback that might improve the TCA treatment? Q7: Are you interested in participating i

CONTACTS AND LOCATIONS:
Overall Officials: Adelaide A Hebert, MD, Principal Investigator — UTHealth McGovern Medical School-Houston and Children's Memorial Hermann Hospital-Houston; Mark J Miller, PhD, Study Director — Miller Biosciences LLC
Locations (1):
- UTHealth McGovern Medical School-Houston and Children's Memorial Hermann Hospital-Houston, 6500 West Loop South, Suite 200-A Texas, Bellaire, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wechter T, Feldman SR, Taylor SL. The Treatment of Primary Focal Hyperhidrosis. Skin Therapy Lett. 2019 Jan;24(1):1-7. PMID 30817880
- [Background] Glaser DA, Hebert A, Pieretti L, Pariser D. Understanding Patient Experience With Hyperhidrosis: A National Survey of 1,985 Patients. J Drugs Dermatol. 2018 Apr 1;17(4):392-396. PMID 29601615